CLINICAL TRIAL: NCT03964740
Title: Effectiveness and Efficiency of Mobile Technology in Disease Control and Healthy Lifestyle Promotion in Asthmatic Overweight/Obese Patients. A Pilot Study.
Brief Title: Effectiveness and Efficiency of Mobile Technology in Disease Control of Asthmatic Obese Patients
Acronym: ASMATIC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI14/01946
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Asthma; Obesity
MeSH Terms: conditions — Asthma; Obesity

STUDY DESIGN:
Intervention Model Description: Single-center open-label controlled pilot study. The interventional group receive a mobile device with an installed application for asthma and obesity control and have protocolized in-person ambulatory visits for asthma and nutrition parameters control while the control study follows a pattern of visits based on the usual clinical practice in the study site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Mobile App intervention group
  Interventions: Other: Mobile App intervention
- Control Group (No Intervention): No intervention group

INTERVENTIONS:
Other: Mobile App intervention — The intervention is based on the interventional group subjects use of a mobile device with an ad-hoc designed application (called ASMATIC). This app permit them (in a daily basis) to record asthma control variables (peak-flow and presence of core symptoms), have daily reminders on their medication for asthma control and decision support for patient disease self-management; and contains advice on healthy lifestyle habits, including personalized diet recommendations based on clinical criteria and associated recipes. The device also permits the study subject to communicate with the hospital and for the study team to review potential issues of interest on the patient's asthma control parameters which might need an intervention such us additional in-person consultations
  Arms: Intervention

SUMMARY:
Single-center open-label randomized pilot study to assess the effectiveness and efficiency of a mobile technology based intervention for asthma and obesity control.

DETAILED DESCRIPTION:
Single-center open-label randomized pilot study to assess the effectiveness and efficiency of a mobile technology based intervention for asthma and obesity control. The interventional group subjects received a mobile device with an ad-hoc designed application (called ASMATIC) which permitted them to record asthma control variables (peak-flow and presence of core symptoms), have daily reminders on their medication for asthma control and advice for healthy lifestyle habits, including personalized diet recommendations and exercise monitoring. The device also permits a bidirectional communication between the patient and the study staff for reporting any emerging issues related to the asthmatic condition of the patient, as the need of additional in-personconsultations. The control group is followed-up based on the study site usual clinical practice, without any specific intervention.

The primary study objective is to evaluate whether the use of the ASMATIC mobile application use improves parameters of asthma control, obesity control, asthma obese patient's quality of life and if it's associated with savings in health-related costs (efficiency assessment), compared to the usual clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. or more.
* Diagnosis of asthma, confirmed by spirometry: positive post bronchodilator test (PBT), defined as an improvement of at least 12% and an increment of at least 200 ml in the absolute value of FEV1 following B-agonist inhalation. In case of negative PBT, asthma diagnoses could be establish if a positive result, defined as a PC20< 8 pgr, was achieved in the Methacholine Challenge Test (MCT).
* BMI of 25 or more.
* Subjects must meet criteria of acceptability of spirometry in at least in three manoeuvres (within a maximun of 8). Acceptability of a spirometry for this protocol purpose is defined by: a) minimum of 6 second exhalation time; b) no cough detected in the first second of expiration; c) 1 second volume plateau.
* Subjects must meet criteria of repeatability of spirometry, defined for this protocol purpose as the three highest accepted FEV1 values to be within 0.10L (100mL) of each other or with a variability of 5% or less.
* Subjects with capacity to handle a smartphone device, with incorporated Android system, and to use and input data on the app ASMATIC, designed for this study purposes.
* Subjects willing to give voluntary, signed informed consent, in accordance with Good Clinical Practice (GCP) guidelines.

Exclusion Criteria:

* Subjects with uncontrolled or severe asthma at study entry, defined by at least one of the following criteria: a) FEV1 <80% of the theorical calculated value and a FEV1/FVC ratio <75% at study entry; b) any severe asthma exacerbation within the two months previous to study entry; c) systemic corticoid or any biological treatment received in the previous 6 months to study entry.
* Any known contraindication for bronchodilator reversibility testing or bronchial provocation tests such us: a) any respiratory tract infection in the previous month to selection; b) pregnancy, lactation or intention to become pregnant during the study; or c) any other contraindication for spirometry found following clinical criteria.
* Subjects with any limitation in their capacity to collaborate and comply with study requirements.
* Active smokers or ex-smokers in the 6 months previous to study entry.
* Subjects currently in immunotherapy treatment or potential candidates for it, including subject suffering a malignant disease.
* Subjects with asthma non controlled risk factors.
* Subjects with any severe or non controlled pathology that compromise their safety during their participation study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in % of Forced Expiratory Volume in the first second (FEV1) from baseline to endpoint | 1 year
  Asthma control assessed through the change in % FEV1 from baseline to endpoint in the interventional group and between the interventional and control groups.

SECONDARY OUTCOMES:
Change in % FEV1 from baseline to weeks 8 and 24. | 6 months
  Asthma control assessed through the change in % FEV1 from baseline to weeks 8 and 24 within the interventional group and between the interventional and control groups.
Change in the Tiffenau index (FEV1/FVC (Forced Vital Capacity) from baseline to endpoint. | 1 year
  Asthma control assessed through the change in the Tiffenau index (FEV1/FVC) from baseline to endpoint in the interventional group and between the interventional and control groups.
Change in the Tiffenau index (FEV1/FVC) from baseline to weeks 8 and 24. | 6 months
  Asthma control assessed through the change in the Tiffenau index (FEV1/FVC) from baseline to weeks 8 and 24 within the interventional group and between the interventional and control groups.
Change in the Body Mass Index (BMI) (measured in kg/m^2) from baseline to endpoint | 1 year
  Change in BMI (measured in kg/m^2) from baseline to endpoint. Comparison within the interventional group and between intervention and control group
Change in abdominal perimeter (measured in cm) from baseline to endpoint | 1 year
  Change in abdominal perimeter (measured in cm) from baseline to endpoint. Comparison within the interventional group and between intervention and control group
Change in neck perimeter (measured in cm) from baseline to endpoint (in male study subjects). | 1 year
  Change in neck perimeter (measured in cm) from baseline to endpoint (in male study subjects). Comparison within the interventional group and between intervention and control group
Change in hip perimeter (measured in cm) from baseline to endpoint (in female study subjects). | 1 year
  Change in hip perimeter (measured in cm) from baseline to endpoint (in female study subjects). Comparison within the interventional group and between intervention and control group
Changes in the Asthma Quality of Life Questionnaire (AQLQ) score from baseline to endpoint | 1 year
  Change in the Asthma Quality of Life Questionnaire (AQLQ) score from baseline to endpoint. AQLQ is a 5-item questionnaire, with a range of scores per item between 0 and 5, and a total range of score range of 0 to 25 points. The comparison is to be made within the interventional group and between intervention and control group.
Change in number of Quality-Adjusted Life Years (QALYs) from baseline to endpoint. | 1 year
  Calculated through the EQ-5D (Euro-Quality of Life Questionnaire of 5 Dimensions) score change from baseline to endpoint. Comparison made between intervention and control group
Healthcare costs of the mean ER consultations related to asthmatic symptoms exacerbation reported by the study subjects during the whole study (measured in euros) | 1 year
  Evaluation of health economic impact of using the mobile app ASMATIC assessed through associated costs of the mean number of visits to ER related to asthmatic symptoms exacerbation reported by the study subjects (measured in euros) during the whole study period in the interventional group vs. the control group. Each consultation in ER has a pre-established cost based on the Andalusian Public Health System standards.
Healthcare costs of Primary Care consultations related to asthmatic symptoms exacerbation reported by the study subjects during the whole study (measured in euros) | 1 year
  Evaluation of health economic impact of using the mobile app ASMATIC assessed through associated costs of the mean number of visits to the Primary Care Physician related to asthmatic symptoms exacerbation reported by the study subjects during the whole study period. Each consultation with the Primary Care Physician has a pre-established cost based on the Andalusian Public Health System standards. Comparison between the interventional group vs. the control group.
Healthcare costs of consultations with the Allergologist (measured in euros) | 1 year
  Evaluation of health economic impact of using the mobile app ASMATIC assessed through associated costs of the mean number of consultations with the Allergologist, measured in euros, during the whole study period in the interventional group vs. the control group. Each consultation with the Allergologist has a pre-established cost based on the Andalusian Public Health System standards.
Total healthcare costs of the consultations in ER, Primary Care and Allergology Service related to the asthmatic condition reported by the patients during the whole study period (measured in euros) | 1 year
  Evaluation of health economic impact of using the mobile app ASMATIC assessed through the associated costs of the mean number of consultations in ER, Primary Care and Allergology Service related to the asthmatic condition reported by the patient during the whole study period (measured in euros). Comparison made in the interventional group vs. the control group. Each consultation in ER, with Primary Care and with the Allergologist has a pre-established cost based on the Andalusian Public Health System standards.
Mean number of days of rescue medication use. | 1 year
  Mean number of days of rescue medication use during the whole study period. The outcome will be evaluated between the interventional and control groups.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Guardia, PhD, MD, Principal Investigator — Service of Allergology. Hospital Universitario Virgen Macarena
Locations (1):
- Service of Allergology. Hospital Universitario Virgen Macarena, Seville, Spain

IPD SHARING:
Plan to Share IPD: No